CLINICAL TRIAL: NCT05029115
Title: The Effect of SGLT-2 Inhibitor in Patient With Atrial Fibrillation and Diabetes Mellitus
Status: Enrolling by invitation | Type: Observational
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BEYOND trial
Record Dates: First submitted 2021-08-22; First posted 2021-08-31 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: SGLT-2 Inhibitor; Atrial Fibrillation; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Atrial Fibrillation; Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SGLT-2 inhibitor administration group: The group who administrated SGLT-2 inhibitor for hypoglycemic medication
  Interventions: Drug: SGLT2 inhibitor
- control: The group who are not administrated SGLT-2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Dapagliflozin, Empagliflozin
  Groups: SGLT-2 inhibitor administration group

SUMMARY:
This study was designed to compare the effects on atrial rhythm control between SGLT2 inhibitor and other oral hypoglycemic agents in patients with atrial fibrillation and diabetes mellitus. We are to compare efficacy and safety between these two groups.

DETAILED DESCRIPTION:
This study is a multicenter, prospective open blinded-endpoint design, 1:1 randomized, and controlled study, with total of 716 patients enrolled from 4-5 centers. The primary outcome is recurrence rate of atrial fibrillation within a year, when recurrence of atrial fibrillation is defined as at least one significant atrial fibrillation documented on 24-hour Holter ECG. Secondary outcomes are atrial fibrillation free survival, atrial fibrillation burden at various time points, ablation rate within a year, atrial fibrillation recurrence rate after ablation within a year, volume of left atrium, NT-ProBNP, Symptom score and Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* At least one episode of atrial fibrillation* that is documented during the prior year by any kind of ECG recording.
* Diabetes mellitus type II was diagnosed. (HBA1c >6.5%) and are using oral hypoglycemic agents only
* At least 20 years old and not older than 80 years old.
* Normal ECG parameters when measured in sinus rhythm (QRS width ≤120 ms, QTc interval <440 ms, and PQ interval ≤210 ms in a 12 lead ECG)
* Able and willing to give informed consent.

Exclusion Criteria:

* Any disease that limits life expectancy under 1 year
* Subject for another clinical trial within the past 2 months
* Under 20 years old or over 80 years old
* Pregnant women
* Lactating women
* Drug abuser
* Type 2 DM treated by recombinant insulin
* Diagnosis of Type 1 DM, MODY, or secondary DM
* HbA1c ≥12% or HbA1c <6.5% at diagnosis
* Previous treatment with any SGLT2 inhibitor
* Renal dysfunction (eGFR-CKD-EPI <30ml/min/1.73m^2)
* Chronic cystitis and/or recurrent genitourinary tract infections (3 or more in the last year)
* Unexplained hematuria at baseline study
* Systolic BP >180mmHg or diastolic BP >100mmHg at baseline study
* Systolic BP <95mmHg at baseline study
* Previous treatment with AF ablation
* Acute cardiovascular event [e.g., stroke, acute coronary syndrome (ACS), revascularization, decompensated HF, sustained ventricular tachycardia, return of spontaneous circulation (ROSC)] <8 weeks prior to baseline study
* Severe valvular disease or have prosthetic valve
* Treatment with chronic oral steroid (>30 consecutive days) at a dose equivalent to oral prednisolone ≥10mg/d, within the past 1 month
* History of any malignancy within 5 years
* Clinically profound hepatic dysfunction
* Clinically uncontrolled thyroid dysfunction
* Patients incapable of completing the trial due to any severe medical condition by clinical decision
* Patients with poor compliance (defined as 80 - 120%), except for reasonable situations judged by physician

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who diagnosed AF and T2DM in one year
Sampling Method: Non-Probability Sample
Enrollment: 716 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
recurrence rate of AF within a year in all participants | during 1 year
  Recurrence rates of AF after stepwise rhythm control therapies including anti-arrhythmic drugs (AAD) and ablation.
recurrence rate of AF within a year in ablated participants | 1 year
  Recurrence rates of AF after stepwise rhythm control therapies including anti-arrhythmic drugs (AAD) and ablation.

SECONDARY OUTCOMES:
Atrial fibrillation free survival | from enrollment to recurrence
  will be compared between two groups as the first of the secondary outcome, analyzed with Kaplan-Meier method and documented on curve
Atrial fibrillation burden | at the enrollment and 3, 6, 9 and 12 months after enrollment
  AF burden is defined as atrial fibrillation time percentage documented on 24-hour Holter ECG
Ablation rate | 1 year
  percentage of patients undergone ablation within a year
Sinus rhythm maintenance rate | at the enrollment and 3, 6, 9 and 12 months after enrollment
  Sinus rhythm is considered stable when either a standard ECG or a 24-hour Holter ECG showed no episode of clinically relevant arrhythmia, including AF, at the time of check-up
Diameter of left atrium | difference between the time of enrollment and the time after 1 year
  mm, measuring by transthoracic echocardiography
NT-proBNP | difference between the time of enrollment and the time after 1 year
  pg/mL
mEHRA (modified European Heart Rhythm Association) symptom score | at the enrollment and 3, 6, 9 and 12 months after enrollment
  1, 2a, 2b, 3 and 4. High score means high AF severity.
Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) score | at the enrollment and after 1 year
  consisted of 20 questions. Lower AFEQT score means high AF severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sumi Jung, Study Director — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha womans university mokdong hospital, Yangcheon, Seoul, South Korea

REFERENCES:
- [Derived] Lee K, Lee SK, Lee J, Jeon BK, Kim TH, Yu HT, Lee JM, Park JK, Baek YS, Kim DH, Shim J, Joung B, Lee MH, Pak HN, Park J. Protocol of BEYOND trial: Clinical BEnefit of sodium-glucose cotransporter-2 (SGLT-2) inhibitors in rhYthm cONtrol of atrial fibrillation in patients with diabetes mellitus. PLoS One. 2023 Jan 18;18(1):e0280359. doi: 10.1371/journal.pone.0280359. eCollection 2023. PMID 36652465